CLINICAL TRIAL: NCT03244540
Title: Efficacy of Regional Analgesia Techniques (Quadratus Lumborum Block and Transversus Abdominis Plane Block) in Acute and Chronic Pain Treatment in Patients After Cesarean Delivery
Brief Title: Regional Analgesia After Cesarean Section
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Lublin (Other)
Responsible Party: Principal Investigator, Michał Borys, associate professor, Medical University of Lublin
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KE-0254/127/2017
Record Dates: First submitted 2017-08-04; First posted 2017-08-09 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Cesarean Section; Pain, Postoperative; Pain, Neuropathic
Keywords: postoperative pain; transversus abdominis plane block; quadratus lumborum block; neuropathic pain
MeSH Terms: conditions — Pain, Postoperative; Neuralgia | interventions — Ropivacaine; Acetaminophen; Analgesia, Patient-Controlled; Dipyrone; Ketoprofen; Bupivacaine

STUDY DESIGN:
Intervention Model Description: Participants were randomized 1:1:1
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants, care providers, and assessors were not aware of type of the block
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PCA (Experimental): Subarchnoid anesthesia with bupivacaine PCA with morphine in the PACU
  Interventions: Drug: Paracetamol; Procedure: subarachnoid anesthesia; Procedure: PCA (patient controlled analgesia); Drug: Metamizol; Drug: Ketoprofen; Drug: Bupivacaine
- TAP (Experimental): Subarchnoid anesthesia with bupivacaine TAP (transversus abdominis plane block) ultrasound-guided regional block between abdominal wall muscles to treat acute postoperative pain. Stimuplex Ultra 360 needle will be used and 0.375 % ropivacaine administered (0.2 mL/kg) at the and of cesarean section.
  PCA with morphine in the PACU
  Interventions: Procedure: TAP (transversus abdominis plane block); Device: Stimuplex Ultra 360 needle; Drug: Ropivacaine; Drug: Paracetamol; Procedure: subarachnoid anesthesia; Procedure: PCA (patient controlled analgesia); Drug: Metamizol; Drug: Ketoprofen; Drug: Bupivacaine
- QLB (Experimental): Subarchnoid anesthesia with bupivacaine QLB (quadratus lumborum block) ultrasound-guided regional block between abdominal wall muscles to treat acute postoperative pain. Stimuplex Ultra 360 needle will be used and 0.375 % ropivacaine administered (0.2 mL/kg) at the and of cesarean section.
  PCA with morphine in the PACU
  Interventions: Procedure: QLB (quadratus lumborum block); Device: Stimuplex Ultra 360 needle; Drug: Ropivacaine; Drug: Paracetamol; Procedure: subarachnoid anesthesia; Procedure: PCA (patient controlled analgesia); Drug: Metamizol; Drug: Ketoprofen; Drug: Bupivacaine

INTERVENTIONS:
Procedure: TAP (transversus abdominis plane block) — ultrasound-guided regional block between abdominal wall muscles to treat acute postoperative pain
  Arms: TAP
Procedure: QLB (quadratus lumborum block) — ultrasound-guided regional block between abdominal wall muscles to treat acute postoperative pain
  Arms: QLB
Device: Stimuplex Ultra 360 needle — ultrasound-guided needle will be used for QLB and TAP and regional blocks
  Arms: QLB; TAP
Drug: Ropivacaine — 0.375 % ropivacaine will be administered for both QLB and TAP (0.2 mL per kg on both sides)
  Arms: QLB; TAP
Drug: Paracetamol — Intravenous paracetamol will be used (1.0 gram), up to 4 grams per day
Procedure: subarachnoid anesthesia — subarachnoid anesthesia for each patients participating in the study with pencil point needle
Procedure: PCA (patient controlled analgesia) — All patients will receive PCA pump with morphine (1 mg/mL, 5 minute interval, no loading dose) after transfer to PACU (post-anesthesia care unit)
Drug: Metamizol — Intravenous metamizol will be used (1.0 gram), up to 4 grams per day
Drug: Ketoprofen — Intravenous ketoprofen will be used (0.1 gram), up to 200 milligrams per day
Drug: Bupivacaine — Subarachnoid anesthesia with spinal bupivacaine (MARCAINE SPINAL 0.5% HEAVY)
  Other Names: Marcaine

SUMMARY:
All patients will be anaesthetized with spinal technique. Each patient will be treated with intravenous morphine - patient controlled analgesia (PCA). 2 of 3 groups of patients will receive ultrasound-guided transversus abdominis plane or quadratus lumborum block to treat postoperative pain. Postoperative pain will measured with visual-analogue scale (VAS). Total morphine consumption and time to the first demand will be noted. 1, 2, 6 months after surgery each patient will be called to assess neuropathic pain with Neuropathic Pain Symptom Inventory (NPSI).

DETAILED DESCRIPTION:
Written consent will be obtained before the cesarean section. Only subarachnoidally anaesthetised patients may participate in the study. Pencil-point spinal needle and bupivacaine (Marcaine Heavy Spinal 0.5 %) will be used.

All patients will receive PCA (patient controlled analgesia) pump with morphine (1 mg/mL, 5 minute interval, no loading dose) after transfer to PACU (post-anesthesia care unit). In PACU vital signs will be monitored.

Each patient will be randomly assigned to one of three groups. In the first group of patients no additional regional analgesia will be performed. In the second and the third group, ultrasound-guided transversus abdominis plane or quadratus lumborum block will be done with 0.375 % ropivacaine (0.2 ml per kg on each side).

Postoperative pain will be measured with VAS (visual-analogue scale) 2, 4, 8, 12 and 24 hours after the end of operation.

Paracetamol, metamizol, ketoprofen may be given as required.

1, 3, 6 months patients will be called to assess neuropathic pain. Neuropathic Pain Symptom Inventory (NPSI) will be used.

ELIGIBILITY:
Inclusion Criteria:

* obtained consent
* singleton pregnancy
* subarachnoid anaesthesia

Exclusion Criteria:

* coagulopathy
* allergy to morphine and local anesthetics
* depression, antidepressant drugs treatment
* epilepsy
* usage of painkiller before surgery
* addiction to alcohol or recreational drugs

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 105 (Actual)
Dates: Start 2017-09-04 (Actual); Primary Completion 2018-10-29 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Postoperative pain measured with VAS | up to 24 hours after surgery
  Acute pain measured with VAS (visual-analogue scale)

SECONDARY OUTCOMES:
Neuropathic pain assessed with NPSI | 6 months from the surgery
  Neuropathic pain occurrence with Neuropathic Pain Symptom Inventory (NPSI)
Morphine consumption | up to 24 hours after surgery
  Total morphine consumption

CONTACTS AND LOCATIONS:
Locations (2):
- Poland (2):
  - Szpital Specjalistyczny PRO-FAMILIA w Rzeszowie, Rzeszów
  - Szpital Kliniczny Dzieciątka Jezus, Warsaw

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kadam VR. Ultrasound-guided quadratus lumborum block as a postoperative analgesic technique for laparotomy. J Anaesthesiol Clin Pharmacol. 2013 Oct;29(4):550-2. doi: 10.4103/0970-9185.119148. PMID 24249997
- [Background] Kadam VR. Ultrasound guided quadratus lumborum block or posterior transversus abdominis plane block catheter infusion as a postoperative analgesic technique for abdominal surgery. J Anaesthesiol Clin Pharmacol. 2015 Jan-Mar;31(1):130-1. doi: 10.4103/0970-9185.150575. No abstract available. PMID 25788791
- [Derived] Borys M, Zamaro A, Horeczy B, Geszka E, Janiak M, Wegrzyn P, Czuczwar M, Piwowarczyk P. Quadratus Lumborum and Transversus Abdominis Plane Blocks and Their Impact on Acute and Chronic Pain in Patients after Cesarean Section: A Randomized Controlled Study. Int J Environ Res Public Health. 2021 Mar 28;18(7):3500. doi: 10.3390/ijerph18073500. PMID 33800559